CLINICAL TRIAL: NCT00907283
Title: Ferrochelating Treatment in Patients Affected by "Neurodegeneration With Brain Iron Accumulation" (NBIA)
Brief Title: Ferrochelating Treatment in Patients Affected by Neurodegeneration With Brain Iron Accumulation (NBIA)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ente Ospedaliero Ospedali Galliera (Other)
Responsible Party: Principal Investigator, Dr. Gian Luca Forni, MD, Ente Ospedaliero Ospedali Galliera
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Deferiprone08; EUDRACT NUMBER 2008-005206-39
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Neurodegenerative Disease; Iron Overload
Keywords: NBIA; Iron overload AND brain; Iron chelation AND neurodegeneration; Brain iron Overload; Neurodegeneration; Brain iron Accumulation
MeSH Terms: conditions — Neurodegenerative Diseases; Iron Overload; Nerve Degeneration | interventions — Deferiprone; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- deferiprone (Experimental): 15 mg/Kg/twice for 1 year
  Interventions: Drug: Deferiprone

INTERVENTIONS:
Drug: Deferiprone — 15 mg/Kg/twice for 1 year
  Other Names: EU/1/99/108/002 Ferriprox 100 mg/ml Oral solution; EU/1/99/108/003 Ferriprox 100 mg/ml Oral solution

SUMMARY:
This trial is a multicenter, unblinded, single-arm pilot study, lasting one year (plus one year extension Amendment n.3 25 August 2009, plus two years follow-up Amendment n.7) , to evaluate the efficacy and safety of the chelator therapy with deferiprone on cerebral iron accumulations. The drug will be administered in the dosage of 15 mg/kg twice daily. The safety and tolerability of the drug will be evaluated by measuring hemochrome every seven days with leukocyte formula count.

At 3, 6 and 12 months from the start of treatment, a neurological evaluation will be performed using several specific evaluation scales (International Cooperative Ataxia Rating Scale (ICARS); Unified Parkinson's Disease Rating Scale (UPDRS); Burke-Fahn-Marsden (BFM)).

Every 6 months of treatment, a brain magnetic resonance image (MRI) aimed at measuring iron overload quantitatively, if possible.

DETAILED DESCRIPTION:
The time interval between Study Start Date and Study First Received was related to bureaucratic problems.

The treatment of systemic iron overload has in recent years improved notably since new drugs and new therapeutic combinations have become available for use. Conversely, therapies for the removal of regional iron overloads on the cerebral level have not been described in the literature.

As it is known, the symptoms resulting from a cerebral iron overload are strongly disabling, reducing the patient's autonomy. Considering that valid therapeutic alternatives of proven preventive and/or curative efficacy in these neurodegenerative diseases do not exist today, the use of lipophilic iron chelators must be considered as a possible therapeutic strategy worthy of deeper study.

Deferiprone is an oral active iron chelator, the use of which is authorized for the treatment of iron overload in patients affected by thalassemia major in conditions of "chelation not suitable for Desferal." In recent years, deferiprone has been applied extensively, demonstrating a good efficacy and tolerability profile.

Unlike deferoxamine, a hydrophilic drug, deferiprone presents chemical-physical characteristics (low molecular weight, favourable octanol:water partition coefficient, neutral charge) that guarantee drug good permeability of mitochondrial walls and the blood-brain barrier.

In a recent study deferiprone (commercial name Ferriprox) was used in 13 patients with Friedreich's ataxia (FA), also treated with idebenone (an experimental drug with an anti-oxidant action), compared with 9 patients affected by FA but treated only with Idebenone. The 9 patients who completed the 6 months of treatment with deferiprone were evaluated from a clinical point of view using the ICARS Scale (International Cooperative Ataxia Rating Score) before the start and after 1 and 6 months of therapy. They also performed a cerebral Magnetic Resonance Imaging before and after 1, 2, 4 and 6 months of treatment. The results were promising. In fact, after 6 months of therapy, a reduction in iron accumulation in specific cerebral areas involved in the pathogenesis of neurodegenerative disease was demonstrated. The patients also presented a significant clinical improvement confirmed by the ICARS score.

Therefore the use of deferiprone, despite the possible side effects (such as gastrointestinal disturbances, a temporary increase in transaminases, and especially agranulocytosis found in about 1% of patients treated with deferiprone), currently represents the only possibility for removing and/or preventing the accumulation of iron in the central nervous system, curing and/or avoiding the most severe and debilitating consequences of a disease for which another therapy does not exist.

The Centers that specialize in the treatment of iron accumulation have acquired significant experience in the use of new oral iron chelators over the last 10 years, which permits deferiprone to be used carefully and safely in the three cases at hand. We therefore propose the use of this drug for treating patients who show neurological symptoms that can be correlated with a cerebral iron overload shown through MRI and who have not benefited from other therapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients over > 1 years of age who have neurological symptoms that can be correlated with cerebral-level iron overload as documented with MRI.This inclusion criteria has been amended by Amendment 6, 24 march 2011)
* Patients who have given informed consent.

Exclusion criteria:

* Inability to be subjected to MRI exam.
* Renal insufficiency (creatinine > 1.5 mg/dl).
* Neoplasias.
* Patients with average levels of ALT > 300 and patients with variations of ALT or AST of 300% during the year prior to enrolling. (At least 4 measurements in 12 months).
* Systemic cardiovascular, renal, hepatic etc., diseases that could counter-indicate the therapeutic options specified.
* Known hypersensitivity to deferiprone.
* Patient judged potentially unreliable and/or uncooperative with regard to study procedures.
* Pregnancy and breastfeeding.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-11; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy and safety of the chelator therapy with deferiprone on cerebral iron accumulations. | 6 months + 6 months (plus one year extension)
  Safety:CBC including ANC will be monitored weekly.If the liver enzymes are greater than 2.5 fold the upper limit of normal, the drug will be withheld and the assessment repeated in 1 week. If the laboratory values continue to be over 2.5 times the upper limit of normal or if the neutrophil counts decrease to less than 1.5 x 109/L (1500 cells/µl) the Patient will be withdrawn from the study. Neutropenia/Agranulocytosis is confirmed as an Absolute Neutrophil Count being less than 1.5 x 109/L (1500 cells/µl) if counts on two consecutive days are both less than 1.5 x 109 (1500 cells/µl).

CONTACTS AND LOCATIONS:
Overall Officials: Gian Luca Forni, MD, Principal Investigator — E.O. Ospedali Galliera. Centro della Microcitemia e delle Anemie Congenite -Ematology - Genoa Italy
Locations (3):
- Italy (3):
  - Neurological Pathology Department, Brotzu Hospital, Cagliari
  - Centre of Microcitemia and Congenital Anemias, Galliera Hospital, Genoa
  - Clinic of Neurology, University of Genoa, Genoa

REFERENCES:
- [Background] Forni GL, Balocco M, Cremonesi L, Abbruzzese G, Parodi RC, Marchese R. Regression of symptoms after selective iron chelation therapy in a case of neurodegeneration with brain iron accumulation. Mov Disord. 2008 Apr 30;23(6):904-7. doi: 10.1002/mds.22002. PMID 18383118
- [Result] Abbruzzese G, Cossu G, Balocco M, Marchese R, Murgia D, Melis M, Galanello R, Barella S, Matta G, Ruffinengo U, Bonuccelli U, Forni GL. A pilot trial of deferiprone for neurodegeneration with brain iron accumulation. Haematologica. 2011 Nov;96(11):1708-11. doi: 10.3324/haematol.2011.043018. Epub 2011 Jul 26. PMID 21791473